CLINICAL TRIAL: NCT03818581
Title: Effect of Suvorexant on Sleep Disturbance in Patients With Chronic Insomnia and Suboptimally Controlled Type 2 Diabetes: A Randomized 3-month Clinical Trial Using a Sequential Parallel Comparison Design
Brief Title: Suvorexant on Sleep Disturbance in Patients With Chronic Insomnia and Suboptimally Controlled Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John Winkelman, MD, PhD, Chief, Sleep Disorders Clinical Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019P000076
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus; Insomnia; Sleep Disorder; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Inflammation | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: Sequential Parallel Comparison Design: subjects will be randomized in a 1:2 ratio to suvorexant 10-20 mg or equivalent placebo for six weeks, followed by re-randomization of placebo non-responders to either suvorexant or placebo in a 1:1 design for six weeks.
Who Masked: Participant, Investigator
Masking Description: The participant, investigator, and clinical research coordinator will remain masked throughout the duration of the study. An unmasked research coordinator will be responsible for assessing mid-point outcomes on the sleep diaries and communicating with the pharmacy for re-randomization medication orders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Group (Active Comparator)
  Interventions: Drug: Suvorexant
- Placebo Responders (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo Non-responders Re-randomized to Treatment (Active Comparator)
  Interventions: Drug: Suvorexant; Other: Placebo
- Placebo Non-responders Re-randomized to Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Suvorexant — 10-mg or 20-mg Suvorexant capsules
  Other Names: Belsomra
  Arms: Placebo Non-responders Re-randomized to Treatment; Treatment Group
Other: Placebo — Matching placebo capsules
  Arms: Placebo Non-responders Re-randomized to Placebo; Placebo Non-responders Re-randomized to Treatment; Placebo Responders

SUMMARY:
The investigators aim to determine the effect of suvorexant on subjective total sleep time (TST) in suboptimally controlled Type 2 diabetics with chronic insomnia in a randomized placebo-controlled trial for 3 months.

DETAILED DESCRIPTION:
Type 2 diabetes results from a progressive insulin secretory defect on the background of insulin resistance and is a growing pandemic and a leading cause of morbidity and mortality. Sleep disturbance is one of the underappreciated and important features of Type 2 diabetes, and may contribute to the development of the disease. In those with established Type 2 diabetes, there is emerging evidence from cross-sectional studies that sleep disturbance affects glycemic control. Although cross-sectional studies suggest a relationship between sleep disturbance and glycemic control in Type 2 diabetes, causality is best investigated by interventional studies. Suvorexant has a comparatively benign side effect profile compared to many of the hypnotic agents typically prescribed for insomnia. The investigators aim to determine the effect of suvorexant on subjective total sleep time (TST), as well as subjective wake after sleep onset, Insomnia Severity Index, HbA1c levels and insulin sensitivity, inflammatory markers, and other subjective sleep endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of any ethnic origin
2. Written informed consent is obtained
3. Speaks and writes in English
4. A willingness and ability to comply with study procedures.
5. Age 25-75 years
6. Diagnosis of Type 2 diabetes with suboptimally controlled blood sugar determined by HbA1c > 6.5% (and < 10.0%) at both the screening and randomization visits
7. No changes in diabetes medication in the previous month
8. DSM-5 criteria for Insomnia Disorder
9. Score on the Insomnia Severity Index (ISI) measure >10, indicating at least a moderate level of insomnia symptoms2
10. Report a total sleep time ≤ 6.5 hours and combined sleep onset latency (SOL) and wake after sleep onset (WASO) > 45 minutes on 7 or more of the 14 nightly sleep logs during both the initial 2-week screening period and the two-week screening run-in period. Combined SOL and WASO does not decrease by more than 50% on the 2-week sleep diary obtained between the screening visit and the randomization visit.

Exclusion Criteria:

1. Sleep and medical factors:

   1. Diagnosis of severe obstructive sleep apnea not using CPAP (can be included if CPAP adherent), or other untreated primary sleep disorders (e.g. narcolepsy, moderate to severe restless legs syndrome)
   2. Shift workers
   3. Use of hypnotic medications more than twice per week in the past month
   4. Unwillingness to not use sedative-hypnotics (other than suvorexant) during the study period
   5. Unwillingness to maintain stable diabetes medication during the study unless medically indicated
   6. Positive urine toxic screen for any drugs of abuse other than marijuana at Screening Visit
   7. HbA1c ≥ 10.0% at either the screening or randomization visit
2. Psychiatric factors:

   1. Current major depressive episode, by report and as indicated by the Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR).
   2. Subjects with active or unstable major psychiatric disorder, who, in the investigator's judgement, require further treatment.
   3. Current alcohol/substance use disorder
3. Medical factors:

   1. Renal or hepatic disease judged to interfere with drug metabolism and excretion
   2. Pregnant or breastfeeding
   3. Malignancy within past 2 years
   4. Surgery within past 3 months
   5. Neurological disorder or cardiovascular disease raising safety concerns about use of suvorexant and/or judged to interfere with ability to assess efficacy of the treatment
   6. Medical instability considered to interfere with study procedures
   7. Concomitant medications with drug interaction or co-administration concerns
   8. Contraindications or allergic responses to suvorexant
   9. History of being treated with suvorexant
4. Lifestyle and other factors:

   1. Travel across two time-zones during the week prior to enrollment
   2. Greater than 6 cups of coffee per day

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Winkelman, MD/PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 108 participants were enrolled. 36 participants did not meet the eligibility criteria post-enrollment, and thus were not randomized. 3 additional participants were removed from the study prior to randomization due to protocol non-adherence. So, a total of 39 participants who were enrolled were not randomized to the study. 69 participants were randomized, but 2 of them were not treated, leaving a total of 67 participants who were treated.
Groups:
- Treatment Group: Suvorexant capsules: 10-mg or 20-mg
- Placebo Non-responders Re-randomized to Treatment: Suvorexant capsules: 10-mg or 20-mg
  Placebo: Matching placebo capsules
- Placebo: Discontinued or withdrew before randomization 2
Period: Overall Study
Arm/Group | Treatment Group | Placebo Responders | Placebo Non-responders Re-randomized to Treatment | Placebo Non-responders Re-randomized to Placebo | Placebo
Started | 23 | 7 | 16 | 18 | 3
Completed | 20 | 7 | 16 | 18 | 0
Not Completed | 3 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Covid-19 | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — No longer met study criteria | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Four participants in the placebo group dropped out before any baseline or follow-up data could be collected. An additional 4 participants in the treatment group dropped out, leaving only 20 participants with interpretable data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Responders | Placebo Non-responders Re-randomized to Treatment | Placebo Non-responders Re-randomized to Placebo | Total
Number analyzed (Participants) | 20 | 7 | 16 | 18 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.5) | 60.6 (7.1) | 61.4 (8.4) | 58.3 (10.1) | 60.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 7 | 12 | 42
  Male | 4 | 0 | 9 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 2 | 5
  Not Hispanic or Latino | 18 | 7 | 15 | 16 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 1 | 0 | 4
  White | 16 | 7 | 14 | 18 | 55
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Subjective Total Sleep Time [Mean (Standard Deviation); unit: Hours] — Subjective Total Sleep Time was measured by asking participants the question: "What was the total amount of sleep that you got last night?"
  This question was asked every day for 2 weeks at baseline. Each participants baseline score was an average of their responses to that question.
  Hours | 5.5 (0.7) | 5.6 (0.9) | 6.3 (0.7) | 6.1 (0.7) | 5.9 (0.8)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index measures insomnia severity on a scale from 0-28, with higher scores indicating worse insomnia severity than lower scores.
  units on a scale | 14.7 (3.2) | 17.3 (3.6) | 17.3 (3.1) | 16.8 (3.8) | 16.1 (3.6)
Wake After Sleep Onset [Mean (Standard Deviation); unit: Minutes] — Wake After Sleep Onset was measured by asking participants the question: "How long were you awake, in total, between the time you fell asleep and before your final awakening?"
  This question was asked every day for 2 weeks at baseline. Each participants baseline score was an average of their responses to that question.
  Minutes | 88.2 (50.7) | 73.8 (41.9) | 64.8 (42.3) | 73.1 (46.7) | 76.1 (44.2)
Calculated Total Sleep Time [Mean (Standard Deviation); unit: Hours] | 6.0 (0.8) | 5.6 (0.9) | 6.4 (0.7) | 6.2 (0.7) | 5.9 (0.8)
Awakenings [Mean (Standard Deviation); unit: Number of Awakenings] | 2.4 (1.0) | 1.5 (0.8) | 2.1 (1.1) | 2.2 (1.2) | 2.1 (0.5)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index measures sleep quality on a scale from 0-21, with higher scores indicating worse sleep quality than lower scores.
  For the purposes of this study, we only used scores from question 6: "During the past month, how would you rate your sleep quality overall?"
  This question is scored from 0-3, with 0 being better sleep quality and 3 being worse sleep quality.
  units on a scale | 1.8 (0.4) | 2.3 (0.8) | 2.1 (0.5) | 2 (0.7) | 2.0 (0.6)
Sleep Onset Latency [Mean (Standard Deviation); unit: Minutes] — Sleep Onset Latency was measured by asking participants the question: "How long did it take you to fall asleep?"
  This question was asked every day for 2 weeks at baseline. Each participants baseline score was an average of their responses to that question.
  Minutes | 35.1 (17.2) | 47.1 (33.7) | 34.9 (26.5) | 29.0 (19.0) | 34.9 (22.5)
Sleep Efficiency [Mean (Standard Deviation); unit: % of time sleeping/time in bed] — Sleep Efficiency is calculated by the following equation: (Total sleep time)/(Time in bed) * 100%
  This information was collected over a 2-week period and then averaged to find each participants baseline score.
  % of time sleeping/time in bed | 75.7 (0.1) | 80.4 (0.03) | 82.9 (0.09) | 80.0 (0.09) | 79.2 (0.09)
Beck's Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — The Beck's Depression Inventory measures depressive symptoms on a scale from 0-63, with higher scores indicating more severe depression than lower scores.
  units on a scale | 8.4 (5.1) | 9.4 (4.6) | 12.1 (8.3) | 9.3 (6.8) | 9.7 (6.4)
Diabetes Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Quality of Life scale measures the quality of life among diabetes patients on a scale from 0-60, with higher scores indicating lower quality of life than lower scores.
  units on a scale | 8.4 (5.1) | 9.4 (4.6) | 12.1 (8.3) | 9.3 (6.8) | 9.7 (6.4)
Diabetes Distress Scale [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Distress scale measures the distress felt by diabetes patients on a scale from 17-102, with higher scores indicating more distress than lower scores.
  units on a scale | 31.9 (13.2) | 34.1 (18.9) | 33 (12.7) | 33.3 (12.4) | 33.3 (13.1)
HbA1c [Mean (Standard Deviation); unit: % of total hemoglobin] | 7.7 (1.0) | 7.5 (0.9) | 7.5 (0.9) | 7.7 (0.7) | 7.6 (0.8)
CRP [Mean (Standard Deviation); unit: mg/L] | 6.5 (8.9) | 8.2 (7.5) | 5.7 (8.3) | 6.0 (10.2) | 6.4 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Total Sleep Time
Description: Total sleep time as reported on daily sleep diaries
Time Frame: 2 weeks
Population: Three participants in the placebo group dropped out before any baseline or follow-up data could be collected. An additional 3 participants in the treatment group dropped out and one participant did not complete the sleep diaries, leaving only 19 participants with interpretable data.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo Non-responders Re-randomized to Treatment: Placebo: Matching placebo capsules
  Suvorexant capsules: 10-mg or 20-mg
Arm/Group | Treatment Group | Placebo Responders | Placebo Non-responders Re-randomized to Treatment | Placebo Non-responders Re-randomized to Placebo
Number analyzed (Participants) | 19 | 7 | 15 | 17
hours | 6.4 (0.8) | 7.0 (0.9) | 6.7 (0.8) | 6.7 (0.7)
Statistical Analysis 1: Comparison: Treatment Group vs Placebo Responders vs Placebo Non-responders Re-randomized to Treatment vs Placebo Non-responders Re-randomized to Placebo; Test type: Superiority; p = 0.15, SPCD analysis

2. Secondary Outcome: Subjective Wake After Sleep Onset
Description: Total time awake after sleep onset as reported on daily sleep diaries
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group | Placebo Responders | Placebo Non-responders Re-randomized to Treatment | Placebo Non-responders Re-randomized to Placebo
Number analyzed (Participants) | 19 | 7 | 14 | 17
minutes | 62.4 (49.6) | 31.4 (21.0) | 36.7 (25.8) | 48.3 (30.6)

3. Secondary Outcome: Insomnia Severity Index
Description: A validated tool to measure insomnia severity, on a scale of 0-28, with a higher score representing greater insomnia severity.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Responders | Placebo Non-responders Re-randomized to Treatment | Placebo Non-responders Re-randomized to Placebo
Number analyzed (Participants) | 19 | 7 | 15 | 17
units on a scale | 7.1 (5.0) | 5.6 (4.1) | 10.9 (5.7) | 9.1 (5.4)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Phase 1 Suvorexant: Suvorexant: 10-mg or 20-mg Suvorexant capsules
  This group includes 22 participants randomized to suvorexant for phase 1. One of the 23 randomized participants was not treated, leaving only 22 with AE data.
- Phase 1 Placebo: Placebo: Matching placebo capsules
  This group includes 43 participants randomized to placebo for phase 1. One of the 44 randomized participants was not treated, leaving only 43 with AE data.
- Phase 2 Suvorexant (From Phase 1 Suvorexant): Suvorexant: 10-mg or 20-mg Suvorexant capsules
  This group includes 20 phase 1 suvorexant participants who continued on suvorexant for phase 2
- Phase 2 Suvorexant (From Phase 1 Placebo Non-Responders): Suvorexant: 10-mg or 20-mg Suvorexant capsules Placebo: Matching placebo capsules
  This group includes 16 phase 1 placebo non-responders re-randomized to suvorexant for phase 2.
- Phase 2 Placebo (From Phase 1 Placebo Non-Responders): Placebo: Matching placebo capsules
  This group includes 18 phase 1 placebo non-responders re-randomized to placebo for phase 2.
- Phase 2 Placebo (From Phase 1 Placebo Responders): Placebo: Matching placebo capsules
  This group includes 7 phase 1 placebo responders who continued on placebo for phase 2.
Arm/Group | Phase 1 Suvorexant | Phase 1 Placebo | Phase 2 Suvorexant (From Phase 1 Suvorexant) | Phase 2 Suvorexant (From Phase 1 Placebo Non-Responders) | Phase 2 Placebo (From Phase 1 Placebo Non-Responders) | Phase 2 Placebo (From Phase 1 Placebo Responders)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/43 | 0/20 | 0/16 | 0/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/43 | 0/20 | 0/16 | 0/18 | 0/7
Other Adverse Events (participants affected / at risk) | 10/22 | 2/43 | 6/20 | 6/16 | 0/18 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Suvorexant (N=22) | Phase 1 Placebo (N=43) | Phase 2 Suvorexant (From Phase 1 Suvorexant) (N=20) | Phase 2 Suvorexant (From Phase 1 Placebo Non-Responders) (N=16) | Phase 2 Placebo (From Phase 1 Placebo Non-Responders) (N=18) | Phase 2 Placebo (From Phase 1 Placebo Responders) (N=7)
Neuropathy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA — Serious case of neuropathy requiring surgical amputation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Suvorexant (N=22) | Phase 1 Placebo (N=43) | Phase 2 Suvorexant (From Phase 1 Suvorexant) (N=20) | Phase 2 Suvorexant (From Phase 1 Placebo Non-Responders) (N=16) | Phase 2 Placebo (From Phase 1 Placebo Non-Responders) (N=18) | Phase 2 Placebo (From Phase 1 Placebo Responders) (N=7)
Grogginess (General disorders) | 5 | 1 | 2 | 3 | 0 | 0
Vivid dreams (General disorders) | 3 | 0 | 1 | 3 | 0 | 1
Headache (General disorders) | 2 | 1 | 1 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03818581/Prot_SAP_000.pdf